CLINICAL TRIAL: NCT06401915
Title: Intelligent Assistive Technologies for Dementia
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Fong Chin Su, Chair Professor, National Cheng-Kung University Hospital
Other Study IDs: B-ER-112-026
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Healthy Adult
Keywords: Dementia Care; Hand rehabilitation; HAAL dashboard

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Platform tester: Participants in this group tested the proposed platform over 6 months, and their feedback were collected 8 times.

SUMMARY:
With the HAAL(HeAlthy Ageing eco system for peopLe with dementia) project, the Netherlands, Taiwan, Italy, Austria, and Denmark combine their strength, co-create, evaluate and share their experiences in supporting dementia care by state-of-the-art AAL bundles.Co-design sessions will take place before developing the dashboard, consisting of (in)formal carers, and older people/clients they care for. The HAAL project will conduct field trials with the first version of the dashboard (Alpha testing) and after Alpha testing, a Beta version of the dashboard will be developed according users' feedback. Then more end-users will be incorporated in Beta testing.The aims of the dashboard are to provide support to reduce the workload of the caregivers and allow psychological relief, which eventually support clients' wellbeing.

ELIGIBILITY:
Inclusion Criteria:

Caregiver

* Principal caregivers of PwD(people with dementia) or organizer or manager of care organization

Care Recipient

* Aged ≥ 65
* Global Deterioration Scale(GDS):2-4 level
* Healthy adult (no skeletal muscle, neurological,eye and hearing disease)

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Tainan city, Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
EQ-5D-5L | 5 minutes
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions.
Zarit Burden Interview | 5 minutes
  The Zarit Caregiver Burden Interview (ZBI) was created by Zarit et al. in 1980 [21]. It is a self-administered instrument composed of 22 items scored on a Likert-type scale with 5 response options: never (0 points), rarely (1 point), sometimes (2 points), quite often (3 points), and almost always (4 points).
The General Anxiety Disorder 7(GAD-7) | 5 minutes
  GAD-7 items reflect the DSM-IV criteria for GAD. Respondents are asked to rate each item for frequency of occurrence using a 4-point Likert scale (Not at all = 0, Several days = 1, More than half the days = 2, and Nearly every day = 3). All responses are summed to calculate the total GAD-7 score.
System Usability Scale | 5 minutes
  Created by John Brooke in 1986, the System Usability Scale (SUS) is a widely used tool for evaluating the usability of software, websites, and other interactive systems. Since then, it has become a standard method for assessing the overall user-friendliness of a product.The System Usability Scale is a Likert Scale which includes 10 questions which users of your website will answer.
  Participants will rank each question from 1 to 5 based on how much they agree with the statement they are reading. 5 means they agree completely, 1 means they disagree vehemently.The average System Usability Scale score is 68. If your score is under 68, then there are probably serious problems with your website usability which you should address. If your score is above 68, then you can relax a little bit.

CONTACTS AND LOCATIONS:
Overall Officials: Fong-Chin Su, Principal Investigator — Chair Professor
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cahill S. WHO's global action plan on the public health response to dementia: some challenges and opportunities. Aging Ment Health. 2020 Feb;24(2):197-199. doi: 10.1080/13607863.2018.1544213. Epub 2019 Jan 2. PMID 30600688
- [Background] Prince M, et al., World Alzheimer Report 2015: The Global Impact of Dementia. 2015: Alzheimer's Disease International.
- [Background] Sun Y, Lee HJ, Yang SC, Chen TF, Lin KN, Lin CC, Wang PN, Tang LY, Chiu MJ. A nationwide survey of mild cognitive impairment and dementia, including very mild dementia, in Taiwan. PLoS One. 2014 Jun 18;9(6):e100303. doi: 10.1371/journal.pone.0100303. eCollection 2014. PMID 24940604
- [Background] Yeh, M.-J., Long-term care system in Taiwan: the 2017 major reform and its challenges. Ageing and Society, 2019. 40(6): p. 1334-1351.
- [Background] Vitaliano PP, Zhang J, Scanlan JM. Is caregiving hazardous to one's physical health? A meta-analysis. Psychol Bull. 2003 Nov;129(6):946-72. doi: 10.1037/0033-2909.129.6.946. PMID 14599289
- [Background] Commission, E.E., Long-Term Care in Ageing Societies-Challenges and Policy Options. 2013, Brussels: European Commission.
- [Background] Reisberg B, Ferris SH, de Leon MJ, Crook T. The Global Deterioration Scale for assessment of primary degenerative dementia. Am J Psychiatry. 1982 Sep;139(9):1136-9. doi: 10.1176/ajp.139.9.1136. PMID 7114305
- [Background] Progression, A.s.P.s. Global Dementia Scale. 2021.
- [Background] Devlin NJ, Krabbe PF. The development of new research methods for the valuation of EQ-5D-5L. Eur J Health Econ. 2013 Jul;14 Suppl 1(Suppl 1):S1-3. doi: 10.1007/s10198-013-0502-3. No abstract available. PMID 23900659
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Ko KT, Yip PK, Liu SI, Huang CR. Chinese version of the Zarit caregiver Burden Interview: a validation study. Am J Geriatr Psychiatry. 2008 Jun;16(6):513-8. doi: 10.1097/JGP.0b013e318167ae5b. PMID 18515696
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Brooke, J., SUS-A quick and dirty usability scale. Usability evaluation in industry, 1996. 189(194): p. 4-7.